CLINICAL TRIAL: NCT00097552
Title: Characterization of Subjects With Turner Syndrome Treated With Growth Hormone in the National Cooperative Growth Study (NCGS)
Brief Title: A Study to Evaluate Subjects With Turner Syndrome Treated With Growth Hormone
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85-036, Substudy 9
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is a multicenter, open-label, observational, postmarketing surveillance study of Genentech growth hormone (GH) products in the treatment of girls with Turner syndrome in the United States and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Are girls with Turner syndrome who are being or will be treated with Nutropin, Nutropin AQ, or Protropin
* Are willing to keep follow-up appointments throughout study participation
* Are girls with Turner syndrome who have submitted Form 4 upon discontinuation and may also submit Form 9

Exclusion Criteria:

* Have Noonan syndrome
* Subjects treated within the last 6 months with a non-Genentech GH preparation
* Have closed epiphyses prior to NCGS enrollment
* Have active neoplasia

Max Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1696 (Actual)
Dates: Start 1997-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lippe, M.D., Study Director — Genentech, Inc.